CLINICAL TRIAL: NCT00657059
Title: A Prospective, Multicenter, Randomized Controlled Trial of Mycophenolate Mofetil (MMF) in Patients With IgA Nephropathy (IgAN)
Brief Title: Mycophenolate Mofetil (MMF) in Patients With IgA Nephropathy (IgAN)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xue Qing Yu, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYSU-PRGIgAN-001
Record Dates: First submitted 2008-04-08; First posted 2008-04-14 (Estimated); Last update posted 2019-12-03 (Actual); Status verified 2019-12

CONDITIONS: IgA Nephropathy
Keywords: IgA nephropathy; mycophenolate mofetil
MeSH Terms: conditions — Glomerulonephritis, IGA | interventions — Irbesartan; Methylprednisolone; Prednisone; prednylidene; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Pred group (Active Comparator): Pred Group: Prednisone treatment Patients will give methylprednisolone intravenously at a dose of 0.5 g/day for 3 days at the start of months 1, 3, and 5; then take oral prednisone (0.5 mg/kg/d) on alternate days. Prednison will be tapered 5 mg per month from the seventh month to the 12th month.
  Interventions: Drug: irbesartan; Drug: methylprednisolone (MP) or prednisone (pred)
- MMF Group (Active Comparator): MMF Group: MMF treatment Patients will take MMF 1.0g bid (wt ≥ 50kg) or 0.75g bid (wt < 50kg) for the first 6-month of drug treatment phase, then 0.5 bid for the remaining 6-month.
  Interventions: Drug: irbesartan; Drug: mycophenolate mofetil (MMF)
- Pred plus MMF Group (Active Comparator): Pred plus MMF Group: Prednisone plus MMF treatment. Patients will give methylprednisolone intravenously at a dose of 0.5 g/day for 3 days at the start of months 1, 3, and 5; then take oral prednisone (0.5 mg/kg/d) on alternate days. Prednison will be tapered 5 mg per month from the seventh month to the 12th month.
  Patients will take MMF 1.0g bid (wt ≥ 50kg) or 0.75g bid (wt < 50kg) for the first 6-month of drug treatment phase, then 0.5 bid for the remaining 6-month.
  Interventions: Drug: irbesartan; Drug: methylprednisolone (MP) or prednisone (pred); Drug: mycophenolate mofetil (MMF)

INTERVENTIONS:
Drug: irbesartan — In the ARB lead-in phase, each subject will be on a strict sodium-restricted diet ( < 5 g NaCl/day), and then given a stable dose (150mg ~ 300mg/day) of irbesartan (Aprovel) for 3 months until reaching the target blood pressure (BP) level of ≤ 125/75 mmHg. Patients will continue ARB treatment in the drug treatment phase and at lease 3 years in the follow-up phase.
  Other Names: Aprovel, Sanofi-synthelabo
Drug: methylprednisolone (MP) or prednisone (pred) — Patients will take oral Pred ( 0.5 mg/kg/d) on alternate days, and on the first, third and fifth months of the drug treatment phase, patients will be given intravenous pulse therapy with methylprednisolone ( 0.5 g/day) for 3 successive days. And after 6 months, Pred should be tapered to be stopped until the end of the 12-month course of treatment.
  Arms: Pred group; Pred plus MMF Group
Drug: mycophenolate mofetil (MMF) — Patients will take MMF 1.0g bid (wt ≥ 50kg) or 0.75g bid (wt < 50kg) for the first 6-month of drug treatment phase, then to 0.5 bid (wt ≥ 50kg) for the remaining 6-month.
  Other Names: Cellcept,Roche
  Arms: MMF Group; Pred plus MMF Group

SUMMARY:
A multi-center, randomized, controlled clinical trial to evaluate the short-term and long-term efficacy and safety of mycophenolate mofetil (MMF) in reducing proteinuria and preserving renal function in patients with IgAN who have pre-treated (and continue to be treated) with angiotensin II receptor blockers (ARB), compared to the corticosteroids.

DETAILED DESCRIPTION:
There are four phases of study for each subject. Phase 1 the screening phase. During this phase each potential subject will be evaluated to determine if he/she is eligible for the study.

Phase 2 the ARB lead-in phase will last for three months. Phase 3 the intervention phase. Each subject will be randomly received 12 months treatment with the study drugs (MMF, prednisone or MMF plus prednisone) Phase 4 following-up phase. All the patients will be followed by 3 years after study drug stopped.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to sign an informed consent
* Age:14~60 years, regardless of gender
* Clinical evaluation and renal biopsy diagnostic for IgAN, excluded secondary IgAN. Renal histological criteria should be defined by Lee's glomerular grading system.
* 1 g/day <= proteinuria < 3.5 g/day, or UPr/Cr ratio ≥ 0.6 (male) or ≥ 0.8 (female) when taking ARB
* eGFR ≥ 40 mL/min/1.73 m2

Exclusion Criteria:

* Inability or unwillingness to sign the informed consent
* Inability or unwillingness to meet the scheme demands raised by the investigators
* Rapidly progressive nephritic syndrome and acute renal failure, including rapidly progressive IgAN ( IgAN with rapid decline in renal function characterized histologically by necrotizing vasculitis and crescent formation≥30%) necessitating the use of other immunosuppressive agents.
* Secondary IgAN such as systemic lupus erythematosus, Henoch-Schonlein purpuric nephritis and hepatitis B -associated nephritis
* est GFR < 40 mL/min/1.73m2
* Malignant hypertension that is difficult to be controlled by oral drugs
* Cirrhosis, chronic active liver disease.
* History of significant gastrointestinal disorders (e.g. severe chronic diarrhea or active peptic ulcer disease.)
* Any Active systemic infection or history of serious infection within one month of entry or known infection with HIV, hepatitis B, or hepatitis C.
* Other major organ system disease (e.g. serious cardiovascular diseases including congestive heart failure , chronic obstructive pulmonary disease, asthma requiring oral steroid treatment or central nervous system diseases)
* Malignant tumors (except fully cured basal cell carcinoma)
* Absolute neutrophil count < 1500／mm3, absolute platelet count <75000／mm3 or hematocrit (Hct) <28% (anemic subjects may be reevaluated after the anemia has been treated.)
* Known allergy, contraindication or intolerance to the MMF, corticosteroids or ACEI/ARB.
* Pregnancy or breast feeding at the time of entry or unwillingness to comply with measures for contraception
* Current exposure to MMF or azathioprine. In case of current treatment with oral steroid or ACEI/ARB, entry is permitted after corticosteroids or ACEI/ARB are stopped for 2 weeks.
* Current or recent (within 30 days) exposure to any other investigational drugs

Ages: 14 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 151 (Actual)
Dates: Start 2007-09; Primary Completion 2019-05 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Remission of proteinuria (complete or partial) | up to 4.3 years

SECONDARY OUTCOMES:
Deterioration of renal function (evidenced by a 50% rise from baseline serum creatinine (SCr) levels, or a 25% decline from baseline eGFR levels, or onset of end-stage renal disease or dialysis treatment, or kidney transplantation) | every 6 month for 4.3 years（including 3 months ARB leading-in phase， 1 years' treatment phase and 3 years' follow-up）

CONTACTS AND LOCATIONS:
Overall Officials: Xueqing Yu, MD, Principal Investigator — Department of Nephrology, 1st Affiliated Hospital, Sun Yat-Sen University; Yunha Liao, MD, Principal Investigator — Department of Nephrology, 1st Affiliated Hospital of Guangxi Medical University,Guangxi; Jinli Zhang, MD, Principal Investigator — Department of nephrology, People's Hospital of Yunnan Province; Junzhou Fu, MD, Principal Investigator — Department of Nephrology,1st People's Hospital of Guangzhou; Anping Xu, MD, Principal Investigator — Department of Nephrology, 2nd Affiliated Hospital of Sun Yet-Sen University,Guangzhou; Zhangsuo liu, MD, Principal Investigator — Department of Nephrology, 1st Affiliated hospital of Zhengzhou University, Henan; Tanqi lou, MD, Principal Investigator — Department of Nephrology, 3nd affiliated hospital of Sun yatsent university, Guangzhou; Li Hao, MD, Principal Investigator — Department of Nephrology, 2nd Affiliated Hospital of Anhui Medical University, Anhui; Menghua Chen, MD, Principal Investigator — Department of Nephrology, General Hospital of Ningxia Medical University, Ningxia; Qinkai Chen, MD, Principal Investigator — Department of Nephrology, The First Affiliated Hospital of Nanchang University, Jiangxi
Locations (1):
- The 1st Affiliated Hospital, Sun Yet-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Alladin A, Hahn D, Hodson EM, Ravani P, Pfister K, Quinn RR, Samuel SM. Immunosuppressive therapy for IgA nephropathy in children. Cochrane Database Syst Rev. 2024 Jun 12;6(6):CD015060. doi: 10.1002/14651858.CD015060.pub2. PMID 38864363